CLINICAL TRIAL: NCT00231010
Title: Molecular Genetics of Retinal Degenerations
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050143; 05-EI-0143
Record Dates: First submitted 2005-09-30; First posted 2005-10-03 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-06-23

CONDITIONS: Retinal Degeneration; Retinitis Pigmentosa
Keywords: Retnitis Pigmentosa; Retinal Degeneration; Retinitis Pigmentosa; RP; Usher Syndrome; USH; Bietti Crystalline Dystrophy; BCD
MeSH Terms: conditions — Retinal Degeneration; Retinitis Pigmentosa; Usher Syndromes; Bietti Crystalline Dystrophy

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other

SUMMARY:
This multinational study will investigate the inheritance of genetic retinal degeneration in families of different nationalities and ethnic backgrounds in order to identify the genes that, when altered, cause retinal degeneration. The retina is a light-sensitive membrane lining the back part of the eye. It relays vision signals to the brain, which the brain interprets into sight. When the retina degenerates, vision is altered and possibly lost. The findings of this study should help improve diagnosis and methods of treatment for these disorders. Participating institutions include: the National Institutes for Health in Bethesda, Maryland; the University of Miami in Florida; the Casey Eye Institute in Portland, Oregon; the Byrd Health Sciences Center in Morgantown, West Virginia; the University of Texas Southwestern Medical School in Dallas, Texas; the University of Tennessee Health Sciences Center in Memphis; the Prasad Eye Institute in Hyderabad, India; National Center of Excellence in Molecular Biology in Lahore, Pakistan; and the Jules Gonin Hospital in Lausanne, Switzerland.

Patients with retinitis pigmentosa and closely related diseases such as Usher syndrome, snowflake vitreoretinal dystrophy and Bietti crystalline dystrophy may be eligible for this study. Participants undergo the following tests and procedures:

* Medical and surgical history, including family history of vision problems.
* Examination to clarify the type of retinal degeneration.
* Eye examination, including tests of color vision, field of vision and ability to see in the dark
* Electroretinogram to test the function of visual cells. For this test, the patient sits in a dark room for 30 minutes with his or her eyes patched. Then, a small electrode (silver disk) is taped to the forehead and the eye patches are removed. The surface the eyes is numbed with eye drops, and contact lenses are placed on the eyes. The patient looks inside a large dark globe that emits a series of light flashes. Then a light is turned on inside the globe and more lights flash. The contact lenses sense small electrical signals generated by the retina when the light flashes.
* Hearing tests for patients with a personal or family history of deafness. Tests include an audiogram, ear examination and test of middle ear function. For middle ear function testing, the patient feels a little air pressure change for a moment and hears some tones. Another test requires the patient to sit quietly with electrodes on the head, forehead and earlobes.
* Balance testing, including walking in a straight line, standing with eyes closed in the dark and other tests of coordination, and caloric testing. For the caloric testing, any ear wax in the ear canal is removed before the test begins. Then, electrodes are placed on the skin near the eyes and on the forehead. A small amount of cool (sometimes cold) or warm water is instilled into each ear canal, first one and then the other.
* Blood sample collection for genetic testing.

DETAILED DESCRIPTION:
Objective: This project, Molecular Genetics of Retinal Degenerations will study the inheritance of genetic retinal degenerations, both Mendelian and complex, in families of many nationalities and ethnic backgrounds in order to identify the genes that, when mutated, cause retinal degenerations and the pathophysiology through which they act.

Study Population: The number of subjects to be enrolled has no logical upper limit, but will be at least 250 and below 5,000 during the next 5 years. The study consists of ascertaining individuals, and especially families with multiple individuals, affected by retinal degenerations including retinitis pigmentosa (RP) and also other closely related retinal degenerations such as Usher syndrome (USH) and Bietti crystalline dystrophy (BCD).

Design: These patients and their families will undergo detailed ophthalmological examinations and, where indicated, additional non-investigational examinations to characterize their retinal degeneration and determine their affectation status. A blood sample will be collected from each individual for isolation of DNA and in some individuals for lymphoblastoid transformation to establish a renewable source of DNA. Linkage analysis, association analysis, physical mapping, and mutational screening will be carried out to identify the specific gene and the mutations in it that are associated with retinal degenerations in this family. If necessary, the gene product will be characterized biochemically.

Outcome Measures: Linkage will be determines using the lod score method and mutations in specific genes will be assessed using a combination of residue conservation, blosum score, and molecular modeling. Association will be determined using chi-square and Fisher exact tests. Biochemical, metabolic, and physiological effects will be individualized to the specific assay.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients that meet diagnostic criteria for specific retinal degenerations will be recruited from the NEI and collaborating clinics.

Subjects with the following will be recruited:

1. Individuals or family members of individuals with Retinal degenerations, either congenital, childhood, or age related.
2. Adults must be capable of providing their own consent.
3. All subjects must be able to cooperate with study examination and phlebotomy.
4. Older than 4 years of age.

EXCLUSION CRITERIA:

1. Diseases, infections, or trauma that mimic primary retinal degenerations.
2. Children requiring sedation for study procedures.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3549 (Actual)
Dates: Start 2005-09-26; Study Completion 2016-06-23

PRIMARY OUTCOMES:
V | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: James F Hejtmancik, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (6):
- United States (3):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Harvard Medical School, Boston, Massachusetts
  - Cleveland Clinic Foundation Childrens Hospital, Cleveland, Ohio
- Sun Yat-Sen University, Guangzhou, China
- Aravind Eye Hospital, Maduri, India
- University of Punjab, Lahore, Pakistan

REFERENCES:
- [Background] Smith RJ, Pelias MZ, Daiger SP, Keats B, Kimberling W, Hejtmancik JF. Clinical variability and genetic heterogeneity within the Acadian Usher population. Am J Med Genet. 1992 Aug 1;43(6):964-9. doi: 10.1002/ajmg.1320430612. PMID 1415347
- [Background] Keats BJ, Todorov AA, Atwood LD, Pelias MZ, Hejtmancik JF, Kimberling WJ, Leppert M, Lewis RA, Smith RJ. Linkage studies of Usher syndrome type 1: exclusion results from the Usher syndrome consortium. Genomics. 1992 Nov;14(3):707-14. doi: 10.1016/s0888-7543(05)80172-7. PMID 1427898
- [Background] Smith RJ, Lee EC, Kimberling WJ, Daiger SP, Pelias MZ, Keats BJ, Jay M, Bird A, Reardon W, Guest M, et al. Localization of two genes for Usher syndrome type I to chromosome 11. Genomics. 1992 Dec;14(4):995-1002. doi: 10.1016/s0888-7543(05)80122-3. PMID 1478678